CLINICAL TRIAL: NCT05477407
Title: A Pathogenesis Pilot Study to Evaluate the Impact of Switching to Tenofovir/lamivudine/doravirine on Adipose Tissue (AT) Morphology and Functions in Suppressed Patients with Weight Gain on an INSTI-based Regimen
Brief Title: Adipose Tissue After Switch to Doravirine
Acronym: ADDORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CREPATS 14
Record Dates: First submitted 2022-07-22; First posted 2022-07-28 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: ADDORE is a pilot, open, single arm pathogenesis study to evaluate the impact on adipose tissue (AT) of a switch to TDF/FTC/DOR at week 48 in 20 patients with a body-weight gain under an INSTI-based regimen (RAL or DTG or BIC) Each patient will be evaluated with an adipose tissue biopsy performed just prior (D0) and after week 48 (W48) of switching from an INSTI-based regimen to a non INSTI-based regimen combining TDF/3TC/Doravirine (Delstrigo®).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pathogenesis study (Experimental): This pathogenesis study aimed to evaluate potential changes in adipose tissue after switching from an INSTI-based regimen (RAL or DTG or BIC) to TDF/FTC/DOR.
  Interventions: Drug: Switch from an INSTI-based regimen to the non INSTI-based regimen combining TDF/3TC/Doravirine

INTERVENTIONS:
Drug: Switch from an INSTI-based regimen to the non INSTI-based regimen combining TDF/3TC/Doravirine — Each patient will be evaluated with an adipose tissue biopsy performed before (D0) and after a 48 week switch (W48) from an INSTI-based regimen to the non INSTI-based regimen combining TDF/3TC/Doravirine (Delstrigo®)

SUMMARY:
Integrase-strand-transfer-inhibitors (INSTIs) based regimens have been associated with body weight gain and increase in total body adipose tissue (AT). Whereas there is by now no clear understanding of the mechanisms that induce these changes, we have observed modifications of AT in vitro, in animals models or in vivo in obese patients with raltegravir (RAL) and dolutegravir (DTG) with the presence of increased peri-adipocyte fibrosis and high levels of collagen VI that have been associated with poor metabolic prognoses together with cellular insulin resistance and decreased adiponectin secretion.

One major clinical question is whether such AT abnormalities are reversible.

Doravirine (DOR), the most recent available Non-Nucleosidic Reverse Transcriptase Inhibitor (NNRTI) drug, has an excellent metabolic profile and as a NNRTI is expected to induce neither changes in fat tissue distribution nor changes in body weight. Tenofovir disoproxil fumarate (TDF) is associated with a protective lipid profile and, unlike tenofovir alafenamide (TAF) which seems to potentiate weight gain in combination with INSTI, has not been associated with weight gain.

One major clinical question is whether such AT abnormalities are reversible.

Doravirine, the most recent available NNRTI drug, has an excellent metabolic profile and as a NNRTI is expected to induce neither changes in fat tissue distribution nor changes in body weight. Tenofovir DF is associated with a protective lipid profile and, unlike TAF which seems to potentiate weight gain in combination with INSTI, has not been associated with weight gain.

We hypothesized that modifications in morphology and function of the adipose tissue in patients with significant weight gain under an INSTI-based regimen could be improved after switching to the triple drug TDF/Emtricitabine/DOR and that fat increase and body weight will be stopped or reversed.

This pathogenesis study aimed to evaluate potential changes in adipose tissue after switching from an INSTI-based regimen (Raltegravir or Dolutegravir or Bictegravir) to TDF/Emtricitabine/DOR. Each patient will be evaluated with an adipose tissue biopsy performed before (D0) and after a 48 week switch (W48) from an INSTI-based regimen to the non INSTI-based regimen combining TDF/3TC/Doravirine.

With a number of 22 patients at D0, a total of 20 patients with paired adipose tissue biopsies are expected at W48.

The antiretroviral therapy with TDF/emtricitabine/Doravirine will be used as routine practice recommends.

DETAILED DESCRIPTION:
Integrase-strand-transfer-inhibitors (INSTIs) represent the most largely prescribed antiretroviral therapy as recommended either as first-line antiretroviral treatment or as switch strategy due to their high efficacy, good tolerability and high genetic barrier to resistance for the latest compounds.

Recently, weight/fat gain has been reported in INSTIs-exposed patients, raising concerns on possible deleterious clinical outcome. Several studies performed in naïve or in Antiretroviral Therapy-suppressed individuals, revealed that dolutegravir (DTG), raltegravir (RAL) or bictegravir (BIC) based therapy resulted in weight gain.

In the large ADVANCE trial, which has compared in Africa three Antiretroviral Therapy initiation strategies, changes in weight, obesity and trunk/limb were greater with dolutegravir/tenofovir alafenamide/Emtricitabine (+6 kg), than with dolutegravir/tenofovir disoproxil fumarate/emtricitabine (+3 kg) and even more than with tenofovir disoproxil fumarate (TDF)/emtricitabine (FTC)/efavirenz (EFV) (+1 kg) at W48.

Women, blacks and persons over 60 years experienced greater weight gain in the two years after versus before switch in the follow-up from 1997-2017 of AIDS-Clinical-Trials-Group (A5001 and A5322) participants who were switched to DTG, RAL or elvitegravir (EVG).

In the Women's Interagency HIV study (WIHS) from 2006-2017, women who switched to or added an INSTI (DTG/RAL/EVG) to Antiretroviral Therapy, experienced mean greater increase in body weight compared to women who did not. The increases in weight gain were limited or not reported in other retrospective studies that included mainly men and Caucasian individuals. However, most of these studies were retrospective and evaluated weight but not fat mass. Reasons for this weight gain are still unknown.

Adipose tissue (AT) plays a major role in the regulation of energy metabolism given its metabolic and secretory functions. In the general population, trunk fat accumulation is associated with alterations in metabolic functions and low-grade inflammation with cardio-metabolic consequences. Adipose tissue inflation disorders such as obesity leads to emergence of fibrosis and low-grade inflammation related to production of pro-inflammatory factors. AT fibrosis is characterized by an impaired remodeling effect on extracellular matrix (ECM) that will limit the " storage capacities" of AT and will favor infiltration by immune cells leading, overall, to a fibro-inflammatory state responsible of several comorbidities such as insulin resistance.

The pathophysiological mechanisms involved in AT dysfunction in the context of HIV infection and INSTI-based treatments are still poorly understood and most likely multifactorial. We recently reported that dolutegravir and raltegravir can directly impact adipocytes and AT and result in higher levels of fibrosis with adipocyte hypertrophy and insulin resistance. Thus, some INSTIs can be responsible for fat gain and associated AT insulin resistance. The possibility that treatment with INSTI could play a role in the onset of diabetes, as suggested by some studies, needs to be further assessed.

Furthermore, recently it has been shown that the "beiging" of AT (presence of beige adipocytes within white AT) exerts a beneficial effect on AT homeostasis. Indeed, these beige adipocytes are characterized by a thermogenic capacity (through the expression of the uncoupling protein UCP1) that favors the increase in energy expenditure and results in a reduction in adipocyte hypertrophy. Interestingly, recent data from the literature suggest that patients receiving INSTIs exhibit a decrease in the expression of "beiging" markers within their subcutaneous AT.

Doravirine (DOR) is a new second generation Non-Nucleosidic Reverse Transcriptase Inhibitor (NNRTI) highly effective both in naïve and experienced patients in combination with tenofovir and lamivudine. It has been shown to be highly effective with no difference in terms of efficacy when compared to the protease inhibitor darunavir or the first generation NNRTI efavirenz. Doravirine is well tolerated with nausea, headache, diarrhea, fatigue, dizziness, abdominal pain, vomiting reported as main doravirine-related adverse event (≥2% incidence).

In terms of metabolic impact, as expected from a NNRTI, doravirine induced significantly less lipid changes compared to boosted darunavir over 96 weeks. In terms of LDL and non-HDL-cholesterol, there was a mean decrease of 4.5 mg/dL in the DOR group compared to a mean increase of 14.0 mg/dL in LDL cholesterol and 17.7 mg/dL in non-HDL cholesterol in the ritonavir-boosted darunavir.

The second large phase III study has compared doravirine 100 mg once daily to efavirenz, a first generation NNRTI, with tenofovir disoproxil fumarate (TDF)/lamivudine (3TC) in the DRIVE-AHEAD study. The rate of suppression with plasma viral load less than 50 copies /ml at week 48, was 84.3% in the DOR/3TC/TDF recipients and 80.8% in the EFV/FTC/TDF group (difference 3.5%, 95% Confidence Interval (CI), -2.0, 9.0). Neurosensorial tolerability, a frequent issue in the NNRTI class, was better with doravirine, with lower rates of dizziness (8.8% vs 37.1%), sleep disorders/disturbances (12.1% vs 25.2%), and altered sensorium (4.4% vs 8.2%) than EFV/FTC/TDF.

There was a benefit for doravirine in terms of changes in LDL-cholesterol (-1.6 vs +8.7 mg/dL) and non-HDL-cholesterol (-3.8 vs +13.3 mg/dL) with DOR/3TC/TDF as compared to EFV/FTC/TDF respectively.

In terms of body weight changes, fat tissue and dual energy x-ray absorptiometry evolution with doravirine, only few data are available. Body weight and Body Mass Index (BMI) have been evaluated in a post-hoc analysis of a phase II 2 and the 2 phase III studies DRIVE Forward and DRIVE Ahead with a total of 855 patients in the DOR groups, 383 in the darunavir group, and 472 in the EFV group. Patients were mostly male (85%), of Caucasian origin (60%) with a median BMI of 25 kg/m2 and body weight of 75 kg. Over 96 weeks, a median body weight increase of 1.5 kg in the DOR groups, 0.7 kg in the darunavir group and 1.0 kg in the EFV group was observed. The rate of patients with >10% weight gain was 14% in the DOR and EFV groups.

In a phase 2 study comparing the combination islatravir/doravirine to TDF/3TC/DOR, no major changes in body weight and body mass index were observed.

Finally, in contrast with all other NNRTIs, One major clinical question is whether such AT abnormalities are reversible; doravirine has no drug-drug interactions, which is a real advantage in patients with metabolic comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive patient > 18 years
* HIV RNA < 50 copies/ml in the last 6 months
* on INSTI based regimen (dual or 3-DR) since at least 6 months
* Creatinine clearance > 60 ml/min
* With a body weight increase defined as:

  * 10% from pre INSTI body weight whatever duration of INSTI duration OR
  * 5% during the first year after INSTI regimen initiation

Exclusion Criteria:

* Prior hypersensitivity to NNRTI
* Resistance to doravirine in past resistance genotype(s) if available
* Full resistance to tenofovir in past resistance genotype(s) if available
* Diabetes, type 1 or type 2 assessed on by fasting glycemia over 7mmol/L, or non-fasting glycemia over 11 mmol/L or receiving anti-diabetic medications.
* Pregnancy and breast feeding
* Prior bariatric surgery
* Hemostasis disorder or hemophilia
* Oral or injectable anti-diabetics, thyroid hormones, growth hormone, insulin, and corticosteroid therapy lasting more than 5 days.
* Body weight increase (in a context of recent tobacco cessation, introduction of psychotropic drugs, corticosteroids for at least one month, dysthyroidism, anabolic treatment or any hormonal therapy 6 months)
* Current antineoplastic chemotherapy
* Patient with instable housing
* Any acute infection or tumor
* Subjects under judicial protection due to temporarily and slightly diminished mental or physical faculties, or under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Measure the phenotype and alterations in adipose tissue to assess the impact of this weight gain | 48 weeks
  Measure the size of adipocytes assessed by Immunohistochemistry experiments Measure the presence of beige adipocytes within the white adipose tissue (Uncoupling protein 1) assessed by Immunohistochemistry experiments Measure the fibrosis (Red Sirius, collagens, fibronectin, Transforming Growth Factor-β, alpha smooth muscle actin) assessed by Immunohistochemistry experiments
Measure of markers of white adipose tissue, brown/beige adipose tissue, to assess changes in gene expression | 48 weeks
  Measure of markers leptin, adiponectin, transforming growth factor beta and fibroblast growth factor 21 assessed by ReverseTranscriptase-Polymerase Chain Reaction
Measure of markers of white adipocytes, brown adipocytes, differentiation lipogenesis, lipolysis enzymes and major players in insulin sensitivity to assess changes in gene expression | 48 weeks
  Measure of markers peroxisome proliferator-activated receptor, enhancer binding protein alpha, Cell death activator CIDE-A, Protein domain containing 16, Peroxisome proliferator-activated receptor gamma coactivator 1-alpha, Uncoupling Protein 1, sterol regulatory element binding protein 1C, hormone-sensitive lipase, ATGL and glucose transport protein 4 assessed by ReverseTranscriptase-Polymerase Chain Reaction
Measure of components of extra cellular matrix to assess changes in gene expression | 48 weeks
  Measure of markers alpha smooth muscle actin, fibronectin, transforming growth factor beta , collagens, connective tissue growth factor, lactate oxidase lipoxygenase assessed by ReverseTranscriptase-Polymerase Chain Reaction

CONTACTS AND LOCATIONS:
Overall Officials: Christine Katlama, MD, Principal Investigator — Pitie Salpetriere Hospital; Valerie Pourcher, MD, Principal Investigator — Pitie Salpetriere Hospital
Locations (1):
- Christine Katlama, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No